CLINICAL TRIAL: NCT03201055
Title: Assessment of Performance, Usability and Acceptance of a Continuous Positive Airway Pressure System to Alleviate Self-reported Snore in Non-apnoeic Participants
Brief Title: Snore Positive Airway Pressure Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: Eden Sleep (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA100517
Record Dates: First submitted 2017-06-22; First posted 2017-06-28 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Non-Apnoeic Snorers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non Apnoeic Snorers (Experimental): Patient's use the Snore Positive airway pressure device for 28 nights.
  Interventions: Device: Snore PAP System

INTERVENTIONS:
Device: Snore PAP System — The Snore PAP system delivers a set Continuous Positive Airway Pressure (CPAP) and consists of a CPAP flow generator and an approved pillows mask.The system will deliver a fixed positive airflow to the participant via approved tubing and pillows mask.

SUMMARY:
This study will aim to assess the acceptance of the Snore PAP system as a treatment concept for snore. The study will subjectively assess participant and bed partner acceptability and usability of the Snore PAP system and objectively assess participant compliance with the Snore PAP system.

ELIGIBILITY:
Inclusion Criteria

* Participants willing to provide written informed consent
* Participants who can read and comprehend written and spoken English
* Participants who are ≥ 18 years of age
* Participants are CPAP naïve
* Participants who are self/ partner reported snorers
* Participants whose ApneaLink study results demonstrate snore
* Participants who are willing to use Nice system in place of current non prescribed methods for alleviating snore
* Participants have a bed partner
* Participant's bed partner willing to answer assessment questionnaire

Exclusion Criteria

* Participants previously diagnosed with obstructive or central sleep apnoea
* Participants whose ApneaLink home study indicates AHI ≥6
* Participants who are pregnant or breastfeeding
* Participants who have a pre-existing lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury)
* Participants with severe bullous lung disease, history of pneumothorax, pathologically low blood pressure, dehydration, cerebrospinal fluid leak, recent cranial surgery or trauma.
* Participants who cannot participate for the duration of the trial
* Participants who are established on bi-level support therapy
* Participants currently using a prescribed medication/ device to alleviate snore
* Participants who are physically unable to comply with the protocol- no access to internet to conduct online visits with researcher or unable to attend clinic for visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Subjectively assess the participant and bed partner acceptability and usability of Snore PAP system | 28 Nights
  Subjective assessment will be assessed using the Likert scale using a 0-10 scale. With 0 being very negative and 10 being very positive.

SECONDARY OUTCOMES:
Subjectively assess the performance of the Snore PAP system in relieving: self-reported and bed partner reported snore in non-apnoeic participants. | 28 Nights
  Subjective assessment will be assessed using the Likert scale using a 0-10 scale. With 0 being very negative and 10 being very positive.
Objectively assess participant compliance with the Snore PAP system | 28 Nights
  Hours used per night

CONTACTS AND LOCATIONS:
Locations (1):
- EdenSleep, New Plymouth, New Zealand

IPD SHARING:
Plan to Share IPD: No